CLINICAL TRIAL: NCT05192811
Title: Evaluation of the Effects of a Probiotic Strain Lactobacillus Paracasei K56 on Body Fat Reduction in Middle-aged Obese Subjects：A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Effect of Intervention With Probiotic K56 on Body Fat Reduction in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Inner Mongolia Yili Industrial Group Co., Ltd (Industry)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210084
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-11

CONDITIONS: Obesity
Keywords: obesity; lactobacillus paracasei; body fat; visceral fat area; gut microbiota
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic K56 (Experimental): Probiotic capsule (lactobacillus paracasei K56 10^9CFU) 1capsule/day , for 60days
  Interventions: Dietary Supplement: Lactobacillus paracasei K56
- placebo (Placebo Comparator): placebo capsule(maltodextrin, 1capsule/day, 60days
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei K56 — probiotic K56 capsule, 1capsule/day (10^9cfu) ,for 60days
  Arms: probiotic K56
Dietary Supplement: placebo — placebo capsule(maltodextrin) , 1capsule/day ,for 60days
  Arms: placebo

SUMMARY:
The aim of the present study was to investigate the effect of intervention with Lactobacillus paracasei K56 on body fat, metabolic risk markers,inflammatory markers and gut microbiota composition in obesity.

DETAILED DESCRIPTION:
Recent data suggest that gut microbiota can function as an environmental factor that modulates the amount of body fat and obese individuals have an altered gut microbiota.The results of previous animal studies have suggest that a probiotic strain Lactobacillus paracasei K56 have reduced high-fat diet induced obesity.

In this randomised,double blind ,placebo controlled study, the participants were randomly assigned to probiotic K56 group or placebo group to evaluate the fat-reducing effect of the Lactobacillus paracasei K56 by continuously supplementing probiotic or placebo capsules.

ELIGIBILITY:
Inclusion Criteria:

* Obesity : BMI>=30kg/m2,or percent body fat(PBF) >=25% for male, >=30% for female.

（Note: If PBF was eligible, it was recommended that 26 ≤ BMI ≤ 40）

* Age: 40 - 65 years old adults
* Who has the conditions to preserve the test samples at low temperature throughout the whole process

Exclusion Criteria:

* Patients with severe chronic diseases（heart, liver, kidney, hematopoietic system, tumor and other serious diseases, mental illness and organ surgery history, etc.) and complications;
* Patients with severe allergy and immunodeficiency;
* Patients with a clear history of gastrointestinal diseases (ulcer, irritable bowel syndrome, etc.);
* History of intervention with fat-reducing drugs or health products in the past 2 months
* Take weight control measures (diet, exercise, etc.) within the past month
* Participation in other clinical trials within the past 3 months
* who have used antibiotics in the past 2weeks ;
* Those who cannot guarantee to maintain their current lifestyle during the trial period
* Those who fail to consume the tested samples as required, or fail to follow up on time, resulting in failure to determine the efficacy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
visceral fat area (cm^2) | 60days
  VFA (cm^2) will be assessed at baseline and after 60days of intervention
percent body fat (%) | 60days
  PBF (%) will be assessed at baseline and after 60days of intervention

SECONDARY OUTCOMES:
body weight | 60days
  Body weight (kg) will be assessed at baseline and after 60days of intervention
Body Mass Index BMI | 60 days
  Body Mass Index (kg/m^2) will be assessed at baseline and after 60days of intervention
waist circumference (cm) | Baseline, 60 days
  will be assessed at baseline and after 60days of intervention
hip circumference(cm) | 60 days
  will be assessed at baseline and after 60days of intervention
waist to hip ratio (WHR) | 60 days
  waist to hip ratio (WHR) will be assessed at baseline and after 60days of intervention
Serum Lipid Profile | 60 days
  Serum total cholesterol(mmol/L)，Serum triglycerides(mmol/L)，Low-density lipoprotein(mmol/L)，High density lipoprotein(mmol/L) will be measured at baseline and after 60days of intervention
fasting blood glucose | 60 days
  fasting blood glucose(mmol/L) will be measured at baseline and after 60days of intervention
Glycated hemoglobin | 60 days
  Glycated hemoglobin(%) will be measured at baseline and after 60days of intervention
Glycosylated albumin | 60days
  Glycosylated albumin(%) will be measured at baseline and after 60days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ying Feng, Ph.D, Study Director — Hua Dong Hospita Affiliated to Fu Dan University, Shanghai,China
Locations (1):
- Hua Dong Hospital Affiliated to Fu Dan University, Shanghai, China